CLINICAL TRIAL: NCT04298151
Title: Clinical Evaluation of Zirconia Reinforced Versus Conventional Viscous Glass Ionomer in Posterior Restorations of Geriatric Patients: Randomized Controlled Trial
Brief Title: Clinical Performance of Zirconia Reinforced GI Versus Conventional Viscous GI in Geriatric Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Doaa Mohammed Mohammed Abdou, Assistant lecturer, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Zirconia GI Conventional GI
Record Dates: First submitted 2020-03-04; First posted 2020-03-06 (Actual); Last update posted 2024-02-06 (Actual); Status verified 2024-02

CONDITIONS: Geriatric; Performance
Keywords: Glass ionomer; Restorations

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- zirconomer improved (Experimental): zirconia reinforced glass ionomer restoration
  Interventions: Drug: Zirconomer Improved
- ketac molar quick aplicap (Active Comparator): conventional viscous glass ionomer restoration
  Interventions: Drug: Ketac Molar quick Aplicap

INTERVENTIONS:
Drug: Zirconomer Improved — glass ionomer restoration reinforced with nano-zirconia particles to improve strength and esthetics
  Other Names: zirconia reinforced GI
  Arms: zirconomer improved
Drug: Ketac Molar quick Aplicap — highly viscous glass ionomer with improved mechanical properties than the conventional GI
  Other Names: KMQ aplicap
  Arms: ketac molar quick aplicap

SUMMARY:
This study is conducted to evaluate the clinical performance of Zirconomer Improved GI restoration compared to Conventional viscous GI restoration in geriatric patients with Posterior carious lesions in class I or II cavities

DETAILED DESCRIPTION:
This study will be conducted to determine the clinical performance of the Zirconia reinforced glass ionomer restorations ( Zirconomer improved) under stress bearing posterior area (class I or claa II cavities) in geriatric population in comparison to Conventional viscous glass ionomer restorations (Ketac molar quick Aplicap) using the modified United States Public Health Service (USPHS) criteria

P: Geriatric Patients with posterior Caries lesions I: Zirconia reinforced GI (Zirconomer Improved) C: Conventional viscous GI, (Ketac Molar quick Aplicap) O: The Clinical performance of the Glass Ionomer restorations Using USPHS Criteria

ELIGIBILITY:
Inclusion Criteria:

* Age range 60-80 years
* Geriatric patients with Class I or II Posterior carious lesions.
* Males or Females.
* Pulp asymptomatic vital carious posterior teeth.
* Co-operative patients approving to participate in the trial.

Exclusion Criteria:

* Age range less than 60 years.
* Disabilities.
* Deep extensive carious cavities that may lead to fracture of the tooth or pulpal affection.
* Teeth with signs and symptoms of irreversible pulpitis or pulp necrosis.
* Heavy smoking.
* Lack of compliance.

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2022-09-01 (Actual); Study Completion 2022-10-01 (Actual)

PRIMARY OUTCOMES:
Clinical performance | 1 year
  clinical performance of the Glass Ionomer restorations using modified USPHS criteria

CONTACTS AND LOCATIONS:
Locations (1):
- Doaa Abdou, Giza, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Klinke T, Daboul A, Turek A, Frankenberger R, Hickel R, Biffar R. Clinical performance during 48 months of two current glass ionomer restorative systems with coatings: a randomized clinical trial in the field. Trials. 2016 May 8;17(1):239. doi: 10.1186/s13063-016-1339-8. PMID 27156000
- [Background] Walia R, Jasuja P, Verma KG, Juneja S, Mathur A, Ahuja L. A comparative evaluation of microleakage and compressive strength of Ketac Molar, Giomer, Zirconomer, and Ceram-x: An in vitro study. J Indian Soc Pedod Prev Dent. 2016 Jul-Sep;34(3):280-4. doi: 10.4103/0970-4388.186746. PMID 27461814
- [Background] Albeshti R, Shahid S. Evaluation of Microleakage in Zirconomer(R): A Zirconia Reinforced Glass Ionomer Cement. Acta Stomatol Croat. 2018 Jun;52(2):97-104. doi: 10.15644/asc52/2/2. PMID 30034008
- [Background] de Franca Lopes CMC, Schubert EW, Martins AS, Loguercio AD, Reis A, Chibinski ACR, Wambier DS. Randomized Clinical Trial of ART Class II Restorations Using Two Glass Ionomer Cements: One-Year Follow-Up. Pediatr Dent. 2018 Mar 15;40(2):98-104. PMID 29663908
- [Background] Friedl K, Hiller KA, Friedl KH. Clinical performance of a new glass ionomer based restoration system: a retrospective cohort study. Dent Mater. 2011 Oct;27(10):1031-7. doi: 10.1016/j.dental.2011.07.004. Epub 2011 Aug 15. PMID 21840585